CLINICAL TRIAL: NCT04464161
Title: The Effects of Perioperative Nutritional Optimization on Blood Markers of Nutritional Status
Brief Title: The Effects of Perioperative Nutritional Optimization on Blood Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-00748
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Intervertebral Disc Disorders With Radiculopathy, Lumbar Region

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): The treatment arm will receive 6 week supply of daily Ensure protein drinks, while the control arm will be instructed to continue their current diet. This includes 2 weeks pre-operatively and 4 weeks post-operatively.
  Interventions: Dietary Supplement: Ensure
- Arm 2 (No Intervention): The control group will be instructed to continue to their regular diets.

INTERVENTIONS:
Dietary Supplement: Ensure — Ensure protein is a complete nutritional drink with 10g, 240 calories, and 27 vitamins and minerals. It is often used as a nutritional supplementation in many hospitals.
  Arms: Arm 1

SUMMARY:
The purpose of this study is to see if taking an oral nutrition supplement (Ensure Nutrition Shake) before and after lumbar spine surgery affects blood tests related the nutritional status of patients. Patients with poor nutritional statuses who undergo elective lumbar spine surgery are at increased risk for complications and longer hospitalizations.

DETAILED DESCRIPTION:
The study will examine whether a simple and cost-effective perioperative nutritional program will affect blood markers of nutritional status (albumin, pre-albumin, transferrin, electrolytes). All patients 55 years and older who are undergoing lumbar spine surgery at our institution by a single surgeon and meet all inclusion criteria will be added to this study. Patients will be randomized into one of two arms; the interventional group will be provide with daily Ensure protein drinks for two weeks pre-operatively and four weeks post-operatively, while the control group will be instructed to continue their current diet plans. Four weeks post-operatively, blood markers (serum albumin, pre-albumin, transferrin, electrolyes) will be obtained to assess objective differences in nutritional status.

N/A

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 55 years and older undergoing primary lumbar spine surgery for the treatment of radiculopathy and other lumbar pathologies
* Patients have the willingness and ability to participate in a study procedure

Exclusion Criteria:

* Patients who are younger than 55 years old
* Patients undergoing revision surgery
* Patients undergoing surgery due to trauma/fractures
* Patients with lactose intolerance

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Difference in blood markers in patients | Baseline, 4 weeks post-operative visit
  Nutritional status of patients undergoing lumbar surgery will be measured by their blood markers. T-tests with a p value of 0.05 will be used for these tests. Chi square and t-tests will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Passias, MD, Principal Investigator — NYU Langone Hleath
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Hesham.saleh@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.